CLINICAL TRIAL: NCT06001112
Title: Immediate Analgesic Effects of Cheek Acupuncture for Acute Gouty Arthritis
Acronym: CAAGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yuping Lin, Clinical Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-06-clinical study
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Acute Gout Arthritis; Acupuncture; Acute Pain
Keywords: Acute Gout Arthritis; acupuncture; Acute pain
MeSH Terms: conditions — Acute Pain | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture group (Experimental): subjects will received cheek acupuncture for one time
  Interventions: Other: cheek acupuncture
- etoricoxib (Active Comparator): subjects will received etoricoxib 120mg for one time
  Interventions: Drug: Etoricoxib

INTERVENTIONS:
Other: cheek acupuncture — Based on the theory of holography and the theory of the Great Sanjiao, the acupoints were chosen under the guidance of the foundation of cheek acupuncture, selecting bilateral Sanjiao acupoints, bilateral head acupoints, foot and ankle acupoints on the affected side, and matching acupuncture points for local strengthening of the foot and ankle acupuncture points, using the triangular needle strengthening method. The treatment was performed with the patient lying on his back in a comfortable position, with routine local disinfection, rapid transdermal needle entry to the acupuncture points, and needle discharge after 30 minutes of needle retention, after which the needle hole was compressed with a cotton ball for a few moments.
  Arms: acupuncture group
Drug: Etoricoxib — etoricoxib 120mg
  Arms: etoricoxib

SUMMARY:
The goal of this clinical trial is to evaluate the immediate analgesic effect and patients' evaluation of the treatment of cheek acupuncture in patients with acute gouty arthritis. The main question it aims to answer are: Does cheek acupuncture has immediate pain relief effects on patients with acute gouty arthritis. Participants will received cheek acupuncture for 30 mins.

If there is a comparison group: Researchers will compare etoricoxib group to see if cheek acupuncture is superior to etoricoxib for improvement of acute pain in subjects with acute gouty arthritis.

DETAILED DESCRIPTION:
The symptoms of acute gouty arthritis (AGA) are extremely painful, but most patients do not begin to experience pain relief until after they have been seen by a doctor and have taken their medication, leaving a time lag between the time they are seen and the time the treatment is effective. In clinical practice, researchers have found that the use of cheek acupuncture at the first visit to the patient often provides some immediate pain relief, but there is no evidence-based evidence for this.

This project was designed as a prospective, randomized, controlled clinical trial, in which patients with AGA who were seen for the first time were studied, and the treatment group was given cheek acupuncture and the control group was given oral etoricoxib tablets. VAS will be recorded before treatment, 0 min, 30 min, 1 h and 2 h after the start of treatment to depict the immediate analgesic efficacy curve and compare the immediate analgesic effect of the two groups at different time points. If the project is successfully completed, it will explore a treatment method for acute gouty arthritis that is fast-acting, painless and effective, eliminating the time lag between consultation and efficacy for the benefit of gout patients.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for acute gouty arthritis and with attacks in the unilateral ankle or first metatarsophalangeal joint;

  * Age ≥18 years old and ≤75 years old, regardless of gender; ③ The gouty arthritis attack is within 48h; ④ Without therapy with targeted topical treatment or self-administered medications including colchicine, anti-inflammatory pain medications, hormones, herbs, etc.

Agreement to comply with the clinician's treatment plan.

Exclusion Criteria:

* Pregnant or breast-feeding

  * Patients with malignant tumors, severe dysfunction of the heart, liver, and kidneys, diabetes mellitus and hypertension

    * Mental disorders that render the patient unable to understand the nature of the study, its scope, and possible outcomes or unable to follow the doctor's advice

      * Allergic to the components of the drug in this study

        * Patients with active peptic ulcers/bleeding, or previous recurrent ulcers/bleeding.

          * History of asthma, urticaria or allergic reactions induced by taking aspirin or other non-steroidal anti-inflammatory drugs

            * Congestive heart failure (New York Heart Association [NYHA] cardiac function class II-IV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scoring (VAS) | baseline, 0 minute, 30 minutes, 1 hour and 2 hours after the start of treatment
  a 10 cm long horizontal or vertical line that divides the pain level into 10 levels (i.e., 1 level for every 1 cm), with the leftmost (or upper) end representing "no pain" and the rightmost (or lower) end representing "severe pain The leftmost (or upper) end represents "no pain" and the rightmost (or lower) end represents "severe pain", and the patient is asked to mark the pain level he/she feels with an "I" on this line.

SECONDARY OUTCOMES:
Patient feedback score | 2 hours after the start of treatment
  an 8-point patient global assessent of treatment response score was used
Immediate pain relief | 2 hours after the start of treatment
  After the efficacy evaluation of the pain index by retesting 2 hours after the first treatment, the degree of pain relief was divided into: immediate efficacy, which means that all the pain was relieved; apparent efficacy, which means that the pain symptoms were significantly relieved; improvement, which means that the pain situation was relieved; and ineffectiveness, which means that the pain was not resolved at all. Immediate apparent efficiency = immediate efficiency + apparent efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Lin, P.D., Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Yupinglin Lin, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
request from the author
Supporting Information: Study Protocol, CSR
Time Frame: 3year after the end of the trial